CLINICAL TRIAL: NCT01551030
Title: Phase II Study of Buparlisib in Metastatic Transitional Cell Carcinoma of the Urothelium
Brief Title: Buparlisib in Metastatic Transitional Cell Carcinoma of the Urothelium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-060
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2020-09

CONDITIONS: Metastatic Transitional Cell Carcinoma of the Urothelium
Keywords: KIDNEY; URETER; URINARY BLADDER; Buparlisib; 11-060
MeSH Terms: interventions — NVP-BKM120

ARMS (1):
- Buparlisib (Experimental): This is an open-label phase II study of the pan-class I selective phosphoinositide 3-kinase (PI3K) inhibitor Buparlisib in patients with metastatic urothelial carcinoma which has progressed despite treatment with prior cytotoxic chemotherapy.
  Interventions: Drug: Buparlisib

INTERVENTIONS:
Drug: Buparlisib — Buparlisib will be administered at a dose of 100 mg orally once daily (two 50 mg capsules) continuously. Intra-patient dose reduction may be required depending on the type and severity of the individual toxicity encountered. Re-staging imaging studies will be performed after every two cycles of treatment (one cycle = 4 weeks). Patients may continue on study as long as they are tolerating therapy and are free of disease progression.

SUMMARY:
The purpose of this study is to learn what effects, good and/or bad, Buparlisib has on advanced urothelial cancer. Buparlisib is a pill that works by shutting down some of the signals in cancer cells that make tumors grow. It is being tested in patients in research studies such as this one. As of 2010, more than 80 patients with various types of cancer have received treatment with Buparlisib in research studies.

This clinical research study is divided into two parts. The goal of the first part of this study is to learn if the study drug Buparlisib can shrink or slow the growth of cancer in patients with urothelial tumors. The goal of the second part of this study is to learn if the study drug Buparlisib can shrink or slow the growth of urothelial tumors in patients known to have certain genetic alterations that cause these types of tumors. The study doctor will inform the patient which part of the study is currently enrolling participants. Participants in both parts of the study will receive the same treatment and tests.

The safety of this drug will also be studied in both parts. The physical state, changes in the size of the tumor, and laboratory findings taken while on-study will help us decide if Buparlisib is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Karnofsky Performance Status (KPS) ≥60%
* Urothelial carcinoma of the bladder, urethra, ureter or renal pelvis, with histologic confirmation at MSKCC. Patients with unresected primary tumors may be enrolled as long as evidence of metastatic disease is also present.
* Patients must have progressive metastatic disease. Progressive disease will be defined as new or progressive lesions on cross-sectional imaging (RECIST Version 1.1).
* Patients must have been previously treated, as defined by the following:

  * Patients must have received treatment with at least one prior cytotoxic chemotherapy agent but not more than four prior cytotoxic chemotherapy agents for urothelial carcinoma. Up to four prior chemotherapy agents are allowed, since conventional chemotherapy ranges from just one drug (e.g., gemcitabine) to regimens that contain four agents (e.g., M-VAC is a four-drug regimen containing methotrexate, vinblastine, doxorubicin, and cisplatin).

The prior therapy must have consisted of at least one of the following: cisplatin, carboplatin, paclitaxel, docetaxel, or gemcitabine.

o The prior cytotoxic agents may have been administered in the perioperative or metastatic setting and may have been administered sequentially (e.g., first-line treatment followed by second-line treatment at time of progression) or as part of a single regimen.

* Patients must have at least one site of measurable disease per RECIST 1.1 criteria that has not been previously irradiated. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation.
* Patients enrolling in the Phase II study must have pre-treatment tumor tissue available for PI3K/Akt pathway marker analysis: One paraffin block, frozen curls or 10 freshly-prepared unstained slides from the most representative single paraffinembedded tumor tissue block should be submitted. Slides from the primary tumor are preferred. If both the primary and metastatic tumor blocks are available, 10 slides from each of the sites should be submitted. If tissue from the primary tumor is not available, a paraffin block or unstained slides from a metastatic site are acceptable. Fine needle aspirates (FNAs) have insufficient tumor tissue and are not permitted.
* Patients enrolling in the Expansion Cohort must have prior mutational testing demonstrating alterations within the PI3K/Akt/mTOR pathway predicted to result in pathway activation.
* Life expectancy of ≥ 12 weeks
* Adequate bone marrow function as shown by: ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L,
* Hemoglobin >9 g/dL
* Total calcium (corrected for serum albumin) within normal limits (bisphosphonate use for malignant hypercalcemia control is not allowed)
* Corrected Calcium = (0.8 * (Normal Albumin - Pt's Albumin)) + Serum Ca
* Potassium and magnesium within normal limits
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within normal range [or ≤ 3.0 x upper limit of normal (ULN) if liver metastases are present]
* Serum bilirubin within normal range (or ≤ 1.5 x ULN if liver metastases are present; or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in patients with welldocumented Gilbert syndrome)
* Serum creatinine ≤ 1.5 x ULN or 24-hour clearance ≥ 50 mL/min
* INR ≤ 2
* Serum amylase and lipase ≤ ULN
* Fasting plasma glucose ≤ 120 mg/dL (6.7 mmol/L)
* Ability to swallow oral medication

Exclusion Criteria:

* Patients who have received prior treatment with a P13K inhibitor.
* Patients receiving any other investigational therapies.
* Patients with a known hypersensitivity to Buparlisib 120 or to its excipients
* Patients with untreated brain metastases are excluded. However, patients may participate in this trial if > 4 weeks from completion of therapy (radiation and/or surgery) for CNS metastases, are clinically stable at the time of registration and are not receiving corticosteroid therapy
* Patients with acute or chronic hepatic or renal disease or pancreatitis
* Patients with the following mood disorders as judged by the Investigator or a psychiatrist, or as a result of patient's mood assessment questionnaire:

  o Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)
* ≥ CTCAE grade 3 anxiety

  o Meet the cut-off score of ≥ 10 in the PHQ-9 or a cut-off of ≥ 15 in the GAD-7 mood scale, respectively, or select a positive response of "1", "2", or "3" to question number 9 regarding the potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9)
* Patients with diarrhea ≥ CTCAE grade 2 or other impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of Buparlisib120 (e.g., ulcerative diseases, uncontrolled, nausea, vomiting, malabsorption syndrome, or small bowel resection)
* Patient has active cardiac disease including any of the following:

Left ventricular ejection fraction (LVEF) < 50% as determined by Multiple Grated acquisition (MUGA) scan or echocardiogram (ECHO)

* QTc > 480 msec on screening ECG (using the QTcF formula)
* Angina pectoris that requires the use of anti-anginal medication
* Ventricular arrhythmias except for benign premature ventricular contractions
* Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
* Conduction abnormality requiring a pacemaker
* Valvular disease with document compromise in cardiac function
* Symptomatic pericarditis

  * Patients with uncontrolled diabetes mellitus or steroid-induced diabetes mellitus.
  * Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
* Significant symptomatic deterioration of lung function. If clinically indicated, pulmonary function tests including measures of lung volumes, DLCO, O2 saturation at rest on room air should be considered to exclude pneumonitis or pulmonary infiltrates

  * Patients who have been treated with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF) ≤ 2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
  * Patients who are currently receiving treatment with any medication that has the potential to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug. Refer to Appendix A for a list of prohibited QT-prolonging medications.

Patients receiving chronic treatment with steroids or another immunosuppressive agent o Note: Topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are allowed. Patients with previously treated brain metastases who are on stable low dose corticosteroid treatment (e.g., dexamethasone 2 mg/day, prednisolone 10 mg/day) for at least 14 days before start of study treatment are eligible.

* Patients who have taken herbal medications and certain fruits within 7 days prior to starting study drug. Herbal medications include, but are not limited to, St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. Fruits include the CYP3A inhibitors Seville oranges, grapefruit, pummelos, or exotic citrus fruits.
* Patients who are currently treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug. Please refer to Appendix A for a list of moderate to strong inhibitors of CYP3A4 (Please note that co-treatment with weak inhibitors of CYP3A4 is allowed).
* Patients who have received chemotherapy or targeted anticancer therapy ≤ 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug or whose side effects from chemotherapy or targeted anticancer therapy have not recovered to a grade 1 before starting the trial.
* Patients who have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) ≤ 5 effective half lives prior to starting study drug or who have not recovered from side effects of such therapy.

Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy

* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug, patients who have not recovered from side effects of any major surgery, or patients who may require major surgery during the course of the study
* Patients who are currently taking therapeutic doses of warfarin sodium or any other coumarin-derivative anticoagulant.

Women who are pregnant or breast feeding or adults of child-bearing potential not employing an effective method of birth control. Women of child-bearing potential, must have a negative serum pregnancy test ≤ 48 hours prior to initiating treatment. Effective methods of birth control.

* Known diagnosis of human immunodeficiency virus (HIV) infection
* History of another malignancy within 3 years, except non-melanoma skin cancer, excised carcinoma in situ of the cervix or adenocarcinoma of the prostate that has been surgically treated with a post-treatment PSA that is non-detectable
* Patients who are unwilling or unable to abide by the study protocol or cooperate fully with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean Bajorin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Buparlisib
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Buparlisib
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 65 [53 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression Free Survival (PFS) at 2 Months
Description: at 2 months for the pan-class I selective PI3K inhibitor Buparlisib in patients with metastatic urothelial cancer that has progressed on prior cytotoxic chemotherapy. Response and progression will be evaluated in this study using the international criteria by the Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: 2 months
Measure: Number; unit: % of participants with PFS
Arm/Group | Buparlisib
Number analyzed (Participants) | 19
% of participants with PFS | 54

2. Primary Outcome: Progression Free Survival (PFS) in the Expansion Cohort
Time Frame: Up to 16 months
Measure: Median (Full Range); unit: months
Arm/Group | Buparlisib
Number analyzed (Participants) | 19
months | 3.2 [1.4 to 15.8]

3. Secondary Outcome: Response Rate
Description: as determined by RECIST v1.1 for Buparlisib in patients with progressive metastatic urothelial cancer who have received prior cytotoxic chemotherapy
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Buparlisib
Number analyzed (Participants) | 19
Participants
  Partial Response | 1
  Stable Disease | 6
  Progression of Disease | 6
  Not Entered | 6

4. Secondary Outcome: Number of Participants Evaluated for Toxicity
Description: To establish the safety and toxicity of Buparlisib , the frequency of toxicity will be tabulated according to the NCI Common Toxicity Criteria, version 4.0.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Buparlisib
Number analyzed (Participants) | 19
Participants | 19

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Buparlisib
All-Cause Mortality (participants affected / at risk) | 17/19
Serious Adverse Events (participants affected / at risk) | 9/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Buparlisib (N=19)
Abdominal pain (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Death NOS (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Platelet count decreased (Investigations) | 1
Sinus tachycardia (Cardiac disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 1
White blood cell decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Buparlisib (N=19)
Fatigue (General disorders) | 15
Hyperglycemia (Metabolism and nutrition disorders) | 15
Weight loss (Investigations) | 11
Alanine aminotransferase increased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 9
Diarrhea (Gastrointestinal disorders) | 7
Mucositis oral (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 7
Dry Skin (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Anemia (Blood and lymphatic system disorders) | 4
Cholesterol high (Investigations) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Photosensitivity (Skin and subcutaneous tissue disorders) | 4
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 4
Activated partial thromboplastin time prolonged (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 3
Anxiety (Psychiatric disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Creatinine increased (Investigations) | 3
Depression (Psychiatric disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 3
Blood bilirubin increased (Investigations) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Edema limbs (General disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Platelet count decreased (Investigations) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Resp, thoracic & mediastinal disorder Other, spec (Respiratory, thoracic and mediastinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Concentration impairment (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
INR increased (Investigations) | 1
Infections and infestations - Other, other (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Rhinitis infective (Infections and infestations) | 1
Stomach pain (Gastrointestinal disorders) | 1
Tremor (Nervous system disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
White blood cell decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT01551030/Prot_SAP_000.pdf